CLINICAL TRIAL: NCT05280444
Title: Transarterial Chemoembolization With Lipiodol-Idarubicin Emulsion in the Treatment of Hepatocellular Carcinoma: a Prospective, Multicenter, Real-world Study
Brief Title: Lipiodol-TACE With Idarubicin for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE-2006
Record Dates: First submitted 2022-03-11; First posted 2022-03-15 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Idarubicin; Real-world study
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Idarubicin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipiodol-TACE with Idarubicin (Experimental): The initial dose of idarubicin is 10 mg and the maximum tolerated dose is 20 mg. Idarubicin is first dissolved in water for injection to make a solvent of 2mg/ml, which is then mixed with lipiodol to make an emulsion with a ratio of 1:2. Lipiodol-idarubicin emulsion is slowly injected, followed by embolization with embolic agents.
  Interventions: Drug: Idarubicin Hydrochloride for Injection

INTERVENTIONS:
Drug: Idarubicin Hydrochloride for Injection — The initial dose of idarubicin is 10 mg and the maximum tolerated dose is 20 mg. Idarubicin is first dissolved in water for injection to make a solvent of 2mg/ml, which is then mixed with lipiodol to make an emulsion with a ratio of 1:2. Lipiodol-idarubicin emulsion is slowly injected, followed by embolization with embolic agents.
  Other Names: Anbijian

SUMMARY:
The purpose of this real-world study is to evaluate the safety and efficacy of lipiodol-TACE with idarubicin for hepatocellular carcinoma.

DETAILED DESCRIPTION:
Idarubicin is a DNA topoisomerase II inhibitor that promotes DNA strand breakage, trapping cells in the G2 phase of the cell cycle and inducing DNA cleavage and cell apoptosis. At the same time, it can be inserted between the DNA base pairs and produce free radicals, thus breaking the DNA double helix structure and inhibiting the extension, replication and transcription of DNA strands. Preclinical studies have shown that idarubicin has higher antitumor activity than epirubicin, especially against SUN-449 human hepatoma cells. In recent years, domestic and foreign scholars have conducted a series of explorations in the treatment of hepatocellular carcinoma with lipiodol-idarubicin emulsion, and have obtained positive results. This proepective， multicenter real-worldstudy aims to evaluate the efficacy and safety of lipiodol-TACE with idarubicin in Chinese HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1).18-75 years old; no gender limit; 2).Confirmed diagnosis of HCC according to histopathology or CNLC guidelines (2019 Edition); 3）Life expectancy≥3 months; 4).Child-Pugh class A or B; 5).ECOG PS of 0 or 1;6).One of the following cases: CNLC stage IIb and IIIa; CNLC stage Ib and IIa patient who is unable or unwilling to receive surgical treatment due to other reasons (such as advanced age, severe liver cirrhosis, etc.); The main portal vein has not been completely obstructed, with abundant collateral vessels, or restore the blood flow by portal vein stent placement; 7). At least one measurable lesion (the length diameter≥10mm); 8).Laboratory indices: WBC≥3.0×109/L; PLT≥50×109/L; Hb≥70g/L; Cr≤1.5×UNL(upper limit of normal); BIL≤2.0×UNL, ALT≤5.0×UNL, AST≤5.0×UNL.

Exclusion Criteria:

1).The coagulation function is severely decreased and cannot be recovered; 2).The main portal vein is completely embolized by cancer embolism, with few collateral vessels; 3).With active hepatitis or severe infection that cannot be treated at the same time; 4). With cachexia or multiple organ failure; 5). With uncontrollable neurological and mental disorders, or poor compliance; 6.) Primary brain tumors or central nervous system metastasis has not been controlled, with obvious intracranial hypertension or neuropsychiatric symptoms; 7). Pregnant or breast feeding women; 8). Received drug treatments in other clinical trial in the past 4 weeks; 9). Other situations where the investigators judge that the patient should not participate in.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) [mRECIST].

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | Up to approximately 2 years
  The DCR is defined as the percentage of participants who have the overall response of CR, PR, or stable disease (SD) [mRECIST].
Time to Progression(TTP) | Up to approximately 2 years
  The TTP is defined as the time from the initiation TACE to tumor progression [mRECIST].
Overall Survival(OS) | Up to approximately 2 years
  The OS is defined as the time from the initiation TACE to death from any cause.
Survival Rate | Up to approximately 2 years
  The proportion of patients who are still alive during the follw-up period.
Adverse Events(AEs) | Up to approximately 2 years
  Incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang A, Hallouch O, Chernyak V, Kamaya A, Sirlin CB. Epidemiology of hepatocellular carcinoma: target population for surveillance and diagnosis. Abdom Radiol (NY). 2018 Jan;43(1):13-25. doi: 10.1007/s00261-017-1209-1. PMID 28647765
- [Result] Bruix J, Gores GJ, Mazzaferro V. Hepatocellular carcinoma: clinical frontiers and perspectives. Gut. 2014 May;63(5):844-55. doi: 10.1136/gutjnl-2013-306627. Epub 2014 Feb 14. PMID 24531850
- [Result] Lencioni R, de Baere T, Soulen MC, Rilling WS, Geschwind JF. Lipiodol transarterial chemoembolization for hepatocellular carcinoma: A systematic review of efficacy and safety data. Hepatology. 2016 Jul;64(1):106-16. doi: 10.1002/hep.28453. Epub 2016 Mar 7. PMID 26765068
- [Result] Pelletier G, Ducreux M, Gay F, Luboinski M, Hagege H, Dao T, Van Steenbergen W, Buffet C, Rougier P, Adler M, Pignon JP, Roche A. Treatment of unresectable hepatocellular carcinoma with lipiodol chemoembolization: a multicenter randomized trial. Groupe CHC. J Hepatol. 1998 Jul;29(1):129-34. doi: 10.1016/s0168-8278(98)80187-6. PMID 9696501
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Camma C, Schepis F, Orlando A, Albanese M, Shahied L, Trevisani F, Andreone P, Craxi A, Cottone M. Transarterial chemoembolization for unresectable hepatocellular carcinoma: meta-analysis of randomized controlled trials. Radiology. 2002 Jul;224(1):47-54. doi: 10.1148/radiol.2241011262. PMID 12091661
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Result] Boulin M, Guiu S, Chauffert B, Aho S, Cercueil JP, Ghiringhelli F, Krause D, Fagnoni P, Hillon P, Bedenne L, Guiu B. Screening of anticancer drugs for chemoembolization of hepatocellular carcinoma. Anticancer Drugs. 2011 Sep;22(8):741-8. doi: 10.1097/CAD.0b013e328346a0c5. PMID 21487286
- [Result] Favelier S, Boulin M, Hamza S, Cercueil JP, Cherblanc V, Lepage C, Hillon P, Chauffert B, Krause D, Guiu B. Lipiodol trans-arterial chemoembolization of hepatocellular carcinoma with idarubicin: first experience. Cardiovasc Intervent Radiol. 2013 Aug;36(4):1039-46. doi: 10.1007/s00270-012-0532-8. Epub 2012 Dec 8. PMID 23224215
- [Result] Tavernier J, Fagnoni P, Chabrot P, Guiu B, Vadot L, Aho S, Boyer L, Abergel A, Hillon P, Sautou V, Boulin M. Comparison of two transarterial chemoembolization strategies for hepatocellular carcinoma. Anticancer Res. 2014 Dec;34(12):7247-53. PMID 25503156
- [Result] Boulin M, Schmitt A, Delhom E, Cercueil JP, Wendremaire M, Imbs DC, Fohlen A, Panaro F, Herrero A, Denys A, Guiu B. Improved stability of lipiodol-drug emulsion for transarterial chemoembolisation of hepatocellular carcinoma results in improved pharmacokinetic profile: Proof of concept using idarubicin. Eur Radiol. 2016 Feb;26(2):601-9. doi: 10.1007/s00330-015-3855-4. Epub 2015 Jun 11. PMID 26060065
- [Result] Guiu B, Jouve JL, Schmitt A, Minello A, Bonnetain F, Cassinotto C, Piron L, Cercueil JP, Loffroy R, Latournerie M, Wendremaire M, Lepage C, Boulin M. Intra-arterial idarubicin_lipiodol without embolisation in hepatocellular carcinoma: The LIDA-B phase I trial. J Hepatol. 2018 Jun;68(6):1163-1171. doi: 10.1016/j.jhep.2018.01.022. Epub 2018 Feb 8. PMID 29427728